CLINICAL TRIAL: NCT03649802
Title: Treating Vitamin D Insufficiency in Community Dwelling Elderly to Improve Arterial Stiffness
Brief Title: Vitamin D and Arterial Stiffness in Elderly
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L18-174
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Vitamin D Deficiency; Arterial Stiffness
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a double blind manner. Arterial stiffness and oxidative stress markers will be evaluated in the low dose Vitamin D (800 IU) versus a high dose vitamin D (5000 IU) over a period of a year
Who Masked: Participant, Investigator
Masking Description: The study coordinators will be aware of the allocation into the low and high dose vitamin D groups but the patient and the investigators will be blinded from this information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low dose Vitamin D-800 IU (Placebo Comparator): Intervention includes low dose arm-800 IU given daily
  Interventions: Dietary Supplement: Low dose vitamin D3
- High dose Vitamin D-5000 IU (Active Comparator): Intervention includes high dose arm-5000 IU given daily
  Interventions: Dietary Supplement: High dose vitamin D3

INTERVENTIONS:
Dietary Supplement: Low dose vitamin D3 — Low dose arm-800 IU given daily
  Arms: Low dose Vitamin D-800 IU
Dietary Supplement: High dose vitamin D3 — High dose arm-5000 IU given daily
  Arms: High dose Vitamin D-5000 IU

SUMMARY:
Investigators will examine arterial stiffness and pulse waveform analysis. Subjects with vitamin D insufficiency will be recruited. A double blind randomized controlled study will examine the effects of standard dose vitamin D3 (800 IU) versus higher dose vitamin D3 (5000 IU)-given on a daily basis.In order to understand mechanisms of action by which vitamin D would improve arterial stiffness investigators will use biomarkers. Oxidative and inflammatory stress will be measured by plasma F2-isoprostanes and Sulforaphane levels.

DETAILED DESCRIPTION:
Cardiovascular disease disproportionately impacts the elderly. Current practice targets vascular disease with aggressive lipid lowering combined with brachial BP regulation, but has only achieved a modest degree of success. There is a need to intervene at a much earlier stage. Increased arterial stiffness is a marker for subclinical vascular disease and a sensitive predictor of ischemic stroke in the elderly. Vitamin D deficiency is linked to an increased risk of vascular disease.

There is an urgent need for well controlled randomized interventional studies in healthy elderly individuals demonstrating that vitamin D levels can improve vascular function in healthy elderly with vitamin D insufficiency. High dose vitamin D (5000 IU) replacement is required to improve systemic inflammation which may contribute to arterial stiffness and vascular aging.

The hypothesis is that daily 5000 IU vitamin D3 will regress or at least prevent progression of arterial stiffness as assessed by the carotid-femoral pulse wave velocity. Furthermore, investigators postulate that this improvement will be linked to improved oxidative and inflammatory status. Investigators will measure plasma measurements of Sulforaphane and plasma F2-isoprostane to assess the anti-oxidative mechanisms by which vitamin D could influence arterial stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling adults (Subjects) aged between 65 and 89 years of age
* Subjects should be ambulatory, living at home and capable of self-care
* Subjects should be able to drive an automobile independently and without assistance
* Subjects agree to home visitation by coordinators to assess pill counts or willing to come to TTUHSC for such a visit every 4 weeks ± 3 days
* 25(OH) Vitamin D value < 30 ng/ml
* Subjects able to read and understand the English language

Exclusion Criteria:

* Subjects unable or unwilling to have follow up for the duration of the study
* Subjects that cannot take a daily Vitamin D supplement or unwilling to have multiple blood draws
* Subjects on peritoneal or hemodialysis or a life expectancy less than 2 years
* Subjects with Sarcoidosis or diseases associated with hypercalcemia
* Subjects with prior cerebrovascular disease or memory problems
* Subjects with prior myocardial infarction or atrial fibrillation or on anticoagulants
* Subjects on medications for memory or cognitive issues or mental health
* Subjects unable to tolerate Sphygamocor and Complior testing protocol

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Carotid-femoral pulse wave velocity measured by equipment provided by Complior pulse wave analysis | 1 year
  Indicator of arterial stiffness meters per second
24 hour BP ambulatory monitoring | 1 year
  Using Central and Brachial BP in mm Hg determination using Sphygmacor
Heart rate variability | 1 year
  Using postural changes to assess heart rate variability in beats per minute using Sphygmacor

SECONDARY OUTCOMES:
Plasma sulphoraphane and F2-isoprostanes. Isoprostanes will be measured by gas chromatography mass spectrometry and sulphoraphane will be measured using LC-MS/MS techniques | 1 year
  Markers for oxidative stress- both markers will be measured in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Pooja N Sethi, MD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States